CLINICAL TRIAL: NCT06333886
Title: Using a Point-of-care Electrophysiological Method to Study the Impact of Neuro-sacral Function on Recovery After Acute Spinal Cord Injuries
Brief Title: Use of Point-of-care Neuro-sacral Electrophysiology Following Spinal Cord Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Andréane Richard-Denis, Associate professor, Department of Medicine, Université de Montréal; Physiatrist, Hôpital du Sacré-Coeur de Montréal; Researcher, CIUSSS du Nord-de-l'Île, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: ciusss-nordmtl_ESG
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries; Neurogenic Bowel; Neurogenic Bladder Dysfunction
Keywords: Spinal cord injury; Electrophysiology; Neuro-sacral dysfunction; Neurogenic bowel and bladder
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCI patients with neuro-sacral dysfunction: 450 patients with traumatic and non-traumatic acute SCI admitted to a level-1 trauma hospital in Montreal, Quebec, Canada
  Interventions: Device: Sacral electromyography

INTERVENTIONS:
Device: Sacral electromyography — Assessment of neuro-sacral function using point-of-care sacral surface electromyography

SUMMARY:
Assessing the sacral nerves is an integral aspect of the evaluation after a spinal cord injury. Being located at the lower end of the spinal cord, the sacral nerves reflect how signals travel through the injured spinal cord. Sacral assessment is therefore essential to determine the level and severity of the spinal cord injury, which helps selecting the proper treatment and predicting recovery (worse when abnormal sacral function. The current assessment relies solely on a manual evaluation, which depends heavily on the physician's experience and does not provide any quantitative value of the dysfunction. The lack of a quantitative method adapted to the clinical setting is a major barrier limiting our knowledge on the impact of sacral function on recovery. We have recently developed an electrophysiological method providing quantitative sacral assessment at bedside after spinal cord injuries. Using this method, we will quantify sacral function in 250 patients with acute spinal cord injuries, and determine its association with recovery 6 months post-injury. We hypothesize that sacral function assessed early within the first 6 weeks after the injury with our method is associated with a better 6-month recovery of motor, sensory, bowel and bladder function. Our objectives are to assess the changes is sacral function during the first 6 months after the injury, and the relationship between early sacral function and 6-month recovery. Sacral function and recovery will be assessed up to 6 months post-injury by the attending physician, in order to measure the electromyographic magnitude of voluntary anal contraction, electromyographic magnitude of anal contraction elicited through sacral reflex testing, and minimal electrical stimulation for which anal sensation is present. The analysis will determine if and how sacral function evolves in time, and if there are specific quantitative criteria of sacral function that physicians can use to determine if patient will have a favorable recovery.

DETAILED DESCRIPTION:
BACKGROUND: Following spinal cord and cauda equina injuries, clinicians perform a neuro-sacral assessment to establish the injury severity, select proper treatment and rehabilitation needs (neuro-sacral dysfunction is an indication for surgery and requires rehabilitation in a specialized facility), and predict recovery. Current assessments rely on a qualitative digital rectal evaluation, which lacks sensitivity and depends heavily on the clinician's experience. Our previous findings suggest that assessing acute neuro-sacral function within the first days post-injury provides important insights on motor, sensory and bowel/bladder recovery. However, the lack of an accessible quantitative evaluation method adapted to the clinical setting is a major barrier limiting our knowledge on neuro-sacral function, hampering the improvement in care management. We have recently validated an quantitative electrophysiological method to assess neuro-sacral function at bedside that preserves the key assessments of the manual evaluation (anal contraction/sensation and sacral reflexes) and eliminates the need to insert the finger into the rectum while being more sensitive to detect changes in neuro-sacral function.

GOALS: We believe that using a quantitative evaluation method is an essential step for optimizing the neurological assessment by clinicians, and for underpinning the impact of early neuro-sacral function on long-term recovery. We therefore hypothesize that acute neuro-sacral function is associated with motor, sensory and bowel/bladder recovery 6 months post-injury.

The specific aims are:

1. Assess longitudinal neuro-sacral function for 6 months post-injury.
2. Assess the relationship between neuro-sacral function and neurofunctional recovery, in order to identify clinical phenotypes of neuro-sacral function and quantitative thresholds associated with improved recovery.

METHODS: For this 4-year longitudinal study, neuro-sacral function and recovery will be assessed in 450 individuals 1, 2, 6 weeks and 6 months after an acute spinal cord and cauda equina injuries. Neuro-sacral assessments will be performed by the attending physiatrist to measure the 1) electromyographic signal amplitude of voluntary anal contraction, 2) electromyographic signal amplitude of anal contraction elicited through anal reflex testing, and 3) perianal electrical perceptual threshold. Study endpoints 6 months post-injury include the improvement in neurological status (primary endpoint: 10-point improvement in motor score) and bowel/bladder function. Longitudinal changes in neuro-sacral function will be characterized from ANOVA. Classification and regression tree analysis will be used to identify clinical phenotypes and objective quantitative thresholds.

EXPECTED OUTCOMES: By implementing an accessible point-of-care quantitative method to assess neuro-sacral function in the clinical setting, we have a real potential to transform the care standards for spinal cord and cauda equina injuries, and improve the efficiency and accuracy for identifying of neuro-sacral dysfunction. We will improve our understanding of the early changes in neuro-sacral dysfunction, therefore bringing new knowledge on the predictors of recovery. We will identify clinical phenotypes of neuro-sacral function and propose objective threshold values to help clinicians identifying proper care trajectory and optimize resources use, using an accessible and validated method that is well tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >/= 18 years
* Spinal cord injury (including cauda equina) due to trauma or extra-dural spinal tumour
* American Spinal Injury Association Impairment Scale grade A, B, C or D
* Neurological level of injury between C0 and S5
* Neurological examination performed prior to surgery according to the ISNCSCI*
* Surgical treatment done at our institution within 5 days of onset of neurological symptoms
* Patient is willing and able to provide informed consent in English or French

Exclusion Criteria:

* Injury not due to blunt trauma or tumour
* Assessment of neuro-sacral function cannot be performed postoperatively within 1 week on the injury (e.g. due to cognitive or brain disorder, sedation, etc.)
* Expected survival less than 6 months
* No spinal surgery performed
* Subacute or chronic spinal cord or cauda equina injury at spinal surgery (delay > 5 days between onset of neurological symptoms and surgery)
* Incomplete or aborted surgical decompression of spinal cord or cauda equina
* Complete spinal cord transection confirmed from preoperative MRI and/or during surgery
* Moderate or severe brain injury (mild traumatic brain injury not an exclusion criteria)
* Associated or preexisting anorectal or pelvic pathology
* Pre-existing neurological disorders such as cerebrovascular disease, Parkinson's disease, multiple sclerosis, stroke, etc.
* Limitation (e.g. in prision, living in another country, unwilling to comply with follow-up visits) to attend follow-up visits up to 6 months after the injury
* Major cognitive deficits precluding informed consent and/or assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute traumatic and atraumatic (tumoral) spinal cord injury patients admitted to a level-1 trauma centre in Montreal, Quebec, Canada requiring spinal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Precise assessment and evaluation of neuro-sacral dysfunction | 4 years
  Improve the precision and accuracy for identifying of neuro-sacral dysfunction and improve understanding of the early changes in neuro-sacral dysfunction, bringing new knowledge on the predictors of recovery. Identification of clinical phenotypes of neuro-sacral function and propose objective threshold values to help clinicians identifying proper care trajectory and optimize resources use, using an accessible and validated method that is well tolerated by patients.

SECONDARY OUTCOMES:
Assessment of clinical phenotypes | 4 years
  Identify clinical phenotypes of neuro-sacral function and propose objective threshold values to better identify individuals with favorable vs. unfavorable neurofunctional recovery
Clinical prognosis assessment | 4 years
  Help clinicians communicate prognosis and select proper care (e.g. define optimal timing for surgery, ideal candidates for specialized rehabilitation, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim V, Mac-Thiong JM, Dionne A, Begin J, Richard-Denis A. Clinical Protocol for Identifying and Managing Bladder Dysfunction during Acute Care after Traumatic Spinal Cord Injury. J Neurotrauma. 2021 Mar 15;38(6):718-724. doi: 10.1089/neu.2020.7190. Epub 2020 Dec 3. PMID 33121377
- [Background] Facchinello Y, Beausejour M, Richard-Denis A, Thompson C, Mac-Thiong JM. Use of Regression Tree Analysis for Predicting the Functional Outcome after Traumatic Spinal Cord Injury. J Neurotrauma. 2021 May 1;38(9):1285-1291. doi: 10.1089/neu.2017.5321. PMID 29065782
- [Background] Kaminski L, Cordemans V, Cernat E, M'Bra KI, Mac-Thiong JM. Functional Outcome Prediction after Traumatic Spinal Cord Injury Based on Acute Clinical Factors. J Neurotrauma. 2017 Jun 15;34(12):2027-2033. doi: 10.1089/neu.2016.4955. Epub 2017 Mar 21. PMID 28129730
- [Background] Denis AR, Feldman D, Thompson C, Mac-Thiong JM. Prediction of functional recovery six months following traumatic spinal cord injury during acute care hospitalization. J Spinal Cord Med. 2018 May;41(3):309-317. doi: 10.1080/10790268.2017.1279818. Epub 2017 Feb 15. PMID 28198660
- [Background] Richard-Denis A, Chatta R, Thompson C, Mac-Thiong JM. Patterns and predictors of functional recovery from the subacute to the chronic phase following a traumatic spinal cord injury: a prospective study. Spinal Cord. 2020 Jan;58(1):43-52. doi: 10.1038/s41393-019-0341-x. Epub 2019 Aug 28. PMID 31462758
- [Background] Richard-Denis A, Beausejour M, Thompson C, Nguyen BH, Mac-Thiong JM. Early Predictors of Global Functional Outcome after Traumatic Spinal Cord Injury: A Systematic Review. J Neurotrauma. 2018 Aug 1;35(15):1705-1725. doi: 10.1089/neu.2017.5403. Epub 2018 Apr 17. PMID 29455634
- [Background] Greciet N, Mac-Thiong JM, Nguyen BH, Richard-Denis A. The Functional Impact of the Absence of a Bulbocavernosus Reflex in the Postoperative Period After a Motor-Complete Traumatic Spinal Cord Injury. Am J Phys Med Rehabil. 2020 Aug;99(8):712-718. doi: 10.1097/PHM.0000000000001398. PMID 32032092
- [Background] Richard-Denis A, Thompson C, Mac-Thiong JM. Quality of life in the subacute period following a cervical traumatic spinal cord injury based on the initial severity of the injury: a prospective cohort study. Spinal Cord. 2018 Nov;56(11):1042-1050. doi: 10.1038/s41393-018-0178-8. Epub 2018 Jul 3. PMID 29970920
- [Background] Richard-Denis A, Benazet D, Thompson C, Mac-Thiong JM. Determining priorities in functional rehabilitation related to quality of life one-year following a traumatic spinal cord injury. J Spinal Cord Med. 2020 Mar;43(2):241-246. doi: 10.1080/10790268.2018.1517138. Epub 2018 Sep 6. PMID 30188803
- [Background] Goulet J, Richard-Denis A, Thompson C, Mac-Thiong JM. Relationships Between Specific Functional Abilities and Health-Related Quality of Life in Chronic Traumatic Spinal Cord Injury. Am J Phys Med Rehabil. 2019 Jan;98(1):14-19. doi: 10.1097/PHM.0000000000001006. PMID 30157080
- [Background] Simpson LA, Eng JJ, Hsieh JT, Wolfe DL; Spinal Cord Injury Rehabilitation Evidence Scire Research Team. The health and life priorities of individuals with spinal cord injury: a systematic review. J Neurotrauma. 2012 May 20;29(8):1548-55. doi: 10.1089/neu.2011.2226. Epub 2012 Apr 18. PMID 22320160
- [Background] Hagen EM. Acute complications of spinal cord injuries. World J Orthop. 2015 Jan 18;6(1):17-23. doi: 10.5312/wjo.v6.i1.17. eCollection 2015 Jan 18. PMID 25621207
- [Background] Fawcett JW, Curt A, Steeves JD, Coleman WP, Tuszynski MH, Lammertse D, Bartlett PF, Blight AR, Dietz V, Ditunno J, Dobkin BH, Havton LA, Ellaway PH, Fehlings MG, Privat A, Grossman R, Guest JD, Kleitman N, Nakamura M, Gaviria M, Short D. Guidelines for the conduct of clinical trials for spinal cord injury as developed by the ICCP panel: spontaneous recovery after spinal cord injury and statistical power needed for therapeutic clinical trials. Spinal Cord. 2007 Mar;45(3):190-205. doi: 10.1038/sj.sc.3102007. Epub 2006 Dec 19. PMID 17179973
- [Background] Kurze I, Geng V, Bothig R. Guideline for the management of neurogenic bowel dysfunction in spinal cord injury/disease. Spinal Cord. 2022 May;60(5):435-443. doi: 10.1038/s41393-022-00786-x. Epub 2022 Mar 25. PMID 35332274
- [Background] Johns J, Krogh K, Rodriguez GM, Eng J, Haller E, Heinen M, Laredo R, Longo W, Montero-Colon W, Wilson C, Korsten M. Management of Neurogenic Bowel Dysfunction in Adults after Spinal Cord Injury: Clinical Practice Guideline for Health Care Providers. Top Spinal Cord Inj Rehabil. 2021 Spring;27(2):75-151. doi: 10.46292/sci2702-75. Epub 2021 May 24. No abstract available. PMID 34108835
- [Background] Gardner A, Gardner E, Morley T. Cauda equina syndrome: a review of the current clinical and medico-legal position. Eur Spine J. 2011 May;20(5):690-7. doi: 10.1007/s00586-010-1668-3. Epub 2010 Dec 31. PMID 21193933